CLINICAL TRIAL: NCT06693791
Title: Efficacy and Safety of a Long-acting Thrombopoietin Receptor Agonist for Platelet Recovery in Adult Hematologic Malignancies Patients Undergoing Umbilical Cord Blood Transplantation
Brief Title: Romiplostim N01 for Platelet Recovery in Adult Hematologic Malignancies Patients Undergoing UCBT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, ph.D, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Romiplostim N01-001
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Platelet Recovery After Umbilical Cord Blood Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Romiplostim N01 (Experimental)
  Interventions: Drug: Romiplostim N01

INTERVENTIONS:
Drug: Romiplostim N01 — Romiplostim N01 was administered subcutaneously once weekly from +1 day to +28 days after UCBT at a recommended starting dose of 5µg/Kg (maximum single dose not to exceed 250µg) for a total of 4 administrations, with the option of continuation of dosing/switching/discontinuing after +28 days, depending on the patient's platelet profile.

SUMMARY:
To evaluate the efficacy and safety of Romiplostim N01 for platelet recovery after umbilical cord blood transplantation (UCBT) in patients with hematological malignancies.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is an important means of curing a wide range of hematologic diseases, and good hematopoietic and immune reconstitution after transplantation is one of the most important factors determining the success of the transplantation.Persistent thrombocytopenia after Allo-HSCT is one of the common post-transplantation complications.This is an investigator-initiated, single-center, single-arm, Phase II clinical trial to evaluate the efficacy and safety of Romiplostim N01 for platelet recovery after UCBT in patients with hematologic tumors. The study was conducted in patients ≥18 years of age with a diagnosis of hematological neoplasia who underwent UCBT. Subjects will be screened and receive roprostin N01 from +1 to +28 days after UCBT after signing an informed consent form, and the study will focus on the cumulative PLT implantation rate at 28 days after transplantation as the primary efficacy measure. The study is planned to enroll 34 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years old, male or female;
* Patients diagnosed with hematological malignancies and undergoing UCBT;
* ECOG score ≤2;
* Voluntary participation in this clinical trial, patients fully understand the trial content and sign the informed consent

Exclusion Criteria:

* Pregnant or lactating women；
* Known allergy to Romiplostim N01;
* A history of severe thrombotic events or known risk factors for thrombosis or active thromboembolism requiring anticoagulation;
* A history of platelet dysfunction or bleeding prone disease or severe bleeding (requiring more than 2 units of red blood cell infusion or a hematocrit drop of ≥10%) within 7 days prior to screening;
* Chronic active hepatitis B and C;
* Repeat or multiple transplantation or multiple organ transplantation;
* HIV positive, EBV-DNA positive, CMV-DNA positive;
* Have severe infection or complicated with serious heart, liver, lung, kidney, neurological or metabolic diseases;
* A serious adverse event (Level 4 or 5) as defined by the Standard General Terminology for Adverse Events Version 4.0 occurred during the pre-treatment period;
* Participants participate in another clinical study with any exploratory drug or device within 30 days prior to baseline visit; Observational studies are allowed;
* Subjects with cognitive impairment or uncontrolled mental illness;
* Subjects and/or authorized family members to refuse treatment with Romiplostim N01;
* Those who are judged by the researchers as not suitable for inclusion (such as accompanying medical history, which may affect the safety of the subjects or it is estimated that the treatment cannot be adhered to due to financial problems).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Time of platelet engraftment | 28 days
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥20 × 10^9/L.
The cumulative incidence of platelet engraftment at 28 days after transplantation | 28 days
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥20 × 10^9/L.

SECONDARY OUTCOMES:
The cumulative incidence of platelet recovery rate at 28 days after transplantation | 28 days
  Platelet recovery was defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥50×10^9/L.
Time of platelet recovery | 28 days
  The Median time of platelet count ≥20×10^9/L, 50×10^9/L, 100×10^9/L without platelet transfusions
Total platelet transfusion during 4 weeks of treatment | 28 days
  Total platelet transfusion during 4 weeks of treatment
Cumulative implantation rate of the granulocyte lineage at 28 days post-transplantation | 28 days
  Absolute neutrophil count (ANC) ≥0.5×10^9/L for 3 consecutive days
Megakaryocyte levels in bone marrow smears 4 weeks after treatment | 4 weeks
  Megakaryocyte levels in bone marrow smears 4 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No